CLINICAL TRIAL: NCT04264689
Title: Perioperative Thoracotomy Analgesia; Different Analgesic Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AP1906-50105
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- thoracic epidural (Active Comparator): thoracic epidural will be done before induction of general anesthesia
  Interventions: Procedure: thoracic epidural
- serratus anterior block (Experimental): ultrasound guided serratus anterior block will be done after induction of general anesthesia
  Interventions: Procedure: serratus anterior block
- erector spinae block (Experimental): ultrasound guided erector spinae block will be done after induction of general anesthesia
  Interventions: Procedure: erector spinae block

INTERVENTIONS:
Procedure: serratus anterior block — ultrasound guided block
  Arms: serratus anterior block
Procedure: thoracic epidural — thoracic epidural
  Arms: thoracic epidural
Procedure: erector spinae block — ultrasound guided block
  Arms: erector spinae block

SUMMARY:
the study aim is to compare the analgesic effect of thoracic epidural versus serratus plane block versus erector spinae block in thoracic surgeries

DETAILED DESCRIPTION:
comparing the analgesic effect of thoracic epidural versus serratus plane block versus erector spinae block in thoracic surgeries regarding pain control and possible side effects

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for thoracotomy age 18-65

Exclusion Criteria:

* patient refusal coagulation defects abnormal kidney or liver functions local infection at site of block bone metastases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
visual analogue score | 24 hours
  minimum value 0 and maximum value 10

SECONDARY OUTCOMES:
mean arterial blood pressure | 24 hours
  measurement of mean arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: walaa Y elsabeeny, MD, Principal Investigator — Lecturer
Locations (1):
- Department of anesthesia and pain medicine. National Cancer Institute, Cairo, Egypt